CLINICAL TRIAL: NCT06167148
Title: Gingival Depigmentation Using Diode Laser 940nm Versus 980nm: A Split-mouth Comparative Clinical Trial
Brief Title: Gingival Depigmentation Using Diode Laser 940nm Versus 980nm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5/23
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Gingival Pigmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 940nm wavelength Diode laser (Experimental)
  Interventions: Device: Biolase Epic X 940nm wavelength Diode laser
- 980nm wavelength Diode laser (Active Comparator)
  Interventions: Device: Doctor smile simpler 980nm wavelength Diode laser

INTERVENTIONS:
Device: Biolase Epic X 940nm wavelength Diode laser — Participants were treated with Biolase Epic X 940nm wavelength Diode laser set at a power of 1 W, fiber 400 µ, irradiation mode: pulsed wave (P3).
  Arms: 940nm wavelength Diode laser
Device: Doctor smile simpler 980nm wavelength Diode laser — Participants were treated with doctor smile simpler 980nm wavelength Diode laser set at a power of 1 W, fiber 400 µ, irradiation mode: pulsed wave (SP).
  Arms: 980nm wavelength Diode laser

SUMMARY:
is study aimed to evaluate the effectiveness of two diode lasers of different wave lengths 940nm and 980nm for the treatment of physiologic gingival melanin hyperpigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes diagnosed clinically with physiologic gingival pigmentation.
* Pigmentation extending from canine to canine in either upper or lower arch.

Exclusion Criteria:

* Smokers.
* Patients with uncontrolled metabolic disease.
* Immuno-compromised patients.
* Patients with renal disease.
* Patients having coagulation disorders.
* Pregnant and lactating women.
* Evidence about the relation of pigmentation with malignancies.
* History of previous treatment of gingival pigmentation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Intensity of pigmentation | up to 12 weeks
  Intensity of pigmentation was assessed with Dummett Oral Pigmentation Index (DOPI 1971).
  DOPI was scored as:
  Score 1: No clinical pigmentation (pink gingiva) Score 2: Mild clinical pigmentation (mild light brown color) Score 3: Moderate clinical pigmentation (medium brown or mixed pink and brown) Score 4: Heavy clinical pigmentation (deep brown or bluish black).
Extension of pigmentation | up to 12 weeks
  Extension of pigmented area was assessed by, Hedin Melanin Index (HMI).
  It was scored as:
  Degree 1: Isolated-only 1 or 2 pigmented interdental papillae Degree 2: Numerous pigmented interdental papillae Degree 3: Short continuous ribbons Degree 4: Long continuous ribbon

CONTACTS AND LOCATIONS:
Overall Officials: Souzy K Anwar, PhD, Principal Investigator — Alexandria University; Yasmine Y Gaweesh, PhD, Study Director — Alexandria University; Nourhan M Aly, MSc, Study Director — Alexandria University; Gillan I El-Kimary, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt